CLINICAL TRIAL: NCT04909840
Title: Effectiveness of the Use of Dental Floss for Gengivite Treatment in Adults: a Randomized Clinical Trial
Brief Title: Effectiveness of the Use of Dental Floss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Carlos Heitor Cunha Moreira, Principal Investigador, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 53831716.5.0000.5346
Record Dates: First submitted 2021-04-12; First posted 2021-06-02 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Gingivitis
Keywords: gingival inflammation; periodontal disease; dental plaque; dental floss
MeSH Terms: conditions — Gingivitis; Periodontal Diseases; Dental Plaque | interventions — Dental Devices, Home Care

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dental floss (Experimental): Instructions of oral hygiene with toothbrush plus dental floss
  Interventions: Other: Instructions oral hygiene with toothbrush plus dental floss
- without dental floss (Active Comparator): Individuals who will use only toothbrush
  Interventions: Other: Instructions oral hygiene with toothbrush only

INTERVENTIONS:
Other: Instructions oral hygiene with toothbrush plus dental floss — Instructions of oral hygiene with toothbrush plus dental floss
  Arms: dental floss
Other: Instructions oral hygiene with toothbrush only — Instructions only with toothbrush
  Arms: without dental floss

SUMMARY:
Bacterial plaque-induced gingivitis is considered the most common oral disease in dentate individuals and the most frequent type of periodontal disease. Manual brushing is the most widely used method for mechanical plaque self-control and, consequently, prevention and treatment of gingivitis. The effectiveness of brushing, however, is questionable in interproximal areas. Thus, interdental cleaning is recognized as an essential part of maintaining gingival health and the most recommended interdental device is dental floss. However, there is weak scientific evidence available about the recommendation for daily flossing. The objective of this randomized blinded trial is to evaluate the efficacy and effectiveness of oral hygiene using soft toothbrush associated with dental floss versus soft toothbrush in maintaining the gingival condition in adults without loss of insertion. Seventy-six subjects with generalized gingivitis at proximal sites will be randomized into two experimental groups according to the use of dental floss: Manual toothbrushing group without the use of dental floss (without dental floss) and Group dental toothbrushing and dental flossing (dental floss). During a period of 8 weeks, the efficacy of the use of the toothbrush associated with the use of the dental floss will be evaluated. After this period, the baseline of the effectiveness study begins. After this period, the baseline of the effectiveness study begins. Participants will be followed up for another 12 months to evaluate the effectiveness of flossing. The parameters Index of Gingival Bleeding (GB) and Plaque Index (PI) will be evaluated at the baseline, 60, 120, 240 and 360 days. Descriptive analysis of GB and PI data will be performed using means, standard deviations and mean percentage of sites with different GB and PI scores. The differences in the means of GB and PI over time between groups and within the same group will be analyzed using the Poisson Multilevel Regression model. The main outcome will be the maintenance of the gingival condition. The difference in interventions will be compared using the chi-square test with significance level of 5%. Adults with less than 15% of sites with gingival bleeding will be considered healthy.

DETAILED DESCRIPTION:
Plaque-induced gingivitis is an inflammation caused by the accumulation of microorganisms around the gingival margins (MARIOTTI, 1999). The bacterial etiology of gingivitis was established by Löe et al. (1965). In this study, the accumulation of plaque on healthy gingiva produced gingivitis between 10 and 21 days and the restitution of oral hygiene procedures for 7 to 10 days reestablished gingival health. Epidemiological data show a high prevalence of gingivitis in the adult population of developed and developing countries (LI et al., 2010; MINISTÉRIO DA SAÚDE, 2011), besides being the most frequent type of periodontal disease (PAGE; BAAB, 1985).

The main clinical outcomes of gingivitis are edema, color change, probing bleeding, increased gingival exudate and sensitivity (PAGE, SCHROEDER, 1976; MARIOTTI, 1999). The clinical signs are restricted to the gingiva and are reversible with the removal of the etiological factor without any damage to the support periodontium (MARIOTTI, 1999). In adition to the local repercussions, the gingival condition has an impact on the quality of life. Self-perception of swollen gums and gingival pain were associated with reduced quality of life (NEEDLEMAN et al., 2004).

Gingivitis is a risk factor in the clinical course of chronic periodontitis. Lang et al. (2009) found that teeth associated with inflamed gingiva had a significantly greater risk of tooth loss than teeth with healthy or slightly inflamed gingiva. Hugoson et al. (2008) showed that improvements in plaque control reduced the prevalence of gingivitis and moderate periodontitis in four cross-sectional studies conducted over 30 years in Sweden. Thus, prevention and treatment of gingivitis can indirectly reduce tooth loss.

The mechanical control of the supragingival plaque is the main mechanism of prevention and treatment of gingivitis (PINTO et al., 2013; SAMBUNJAK et al., 2011). The benefits of adequate plaque control include maintaining a functional dentition, optimizing aesthetic values such as appearance and good breath, reducing the risk of loss of periodontal attachment, and the need for complex, uncomfortable, and costly periodontal treatment (CLAYDON, 2008). In addition, the improvement in periodontal clinical indicators is correlated with an increase in quality of life related to oral health in adults (SHANBHAG; DAHIYA; CROUCHER, 2013).

Manual brushing is the most commonly used method for plaque control. (VAN DER WEIJDEIN; SLOT, 2015). The effectiveness of this procedure depends on the individual ability to remove plaque and the frequency at which this removal is performed (JEPSEN, 1998). The XI European Workshop of Periodontology recommended the daily brushing twice daily with the use of fluoride dentifrice (CHAPPLE et al., 2015). However, Pinto et al. (2013) demonstrated that mechanical self-control with 24-hour frequency is able to prevent gingivitis in subjects with no history of periodontitis. A systematic review showed that a single brushing exercise reduces plaque levels by approximately 42% (SLOT et al., 2012). Randomized clinical trials (ROSEMA et al., 2008; SCHIFF et al., 2006; SHARMA et al., 2002) have shown that manual brushing without the aid of interdental plaque removal devices reduces plaque and gingivitis levels and maintains gingival health.

The effectiveness of brushing, however, is questionable in interproximal areas. In these areas, due to the presence of apical fibers at the point of contact between two adjacent teeth, there is a difficulty of access of dental brushes, which may allow the establishment and maturation of plaque. (SALZER et al., 2015). Thus, removal of interdental plaques is recognized as an essential part of maintaining gingival health (AMERICAN DENTAL ASSOCIATION, 2016; CHAPPLE et al., 2015).

The daily use of dental floss is the recommended procedure for the removal of interdental plaque from areas with papilla filling all interproximal space (AMERICAN DENTAL ASSOCIATION, 2016). However, there is no scientific support for this recommendation. Systematic reviews evaluated the effect of dental floss combined with brushing (BERCHIER et al., 2008; SAMBUNJAK et al., 2011). Berchier et al. (2008) showed that the use of dental floss does not have an additional effect on toothbrushing indices and gingival bleeding. Sambunjak et al. (2011) reported a statistically significant benefit of combined dental floss with tooth brushing only on the reduction of gingivitis in up to 6 months of follow-up. A meta-analysis of these studies concluded that there is poor evidence to support the use of dental floss (SÄLZER et al., 2015).

The evaluation of the effectiveness of interdental cleaning methods should consider the efficacy, acceptability and adherence of the individual to the method (ASADOORIAN; LOCKER, 2006; WARREN; CHATER, 1996). Regular dental use among adults is low (ASADOORIAN & LOCKER, 2006; RIMONDINI et al., 2001; SCHUZ et al., 2006) due to lack of individual ability and motivation (ASADOORIAN; LOCKER, 2006; TEDESCO, KEFFER; FLECK-KANDATH, 1991). Schüz et al. (2009) tested the effect of a behavioral intervention on flossing. The authors concluded that the individual incentive to form a detailed plan on when, where and how to use dental floss, significantly improved their frequency of use.

Therefore, there is weak scientific evidence available regarding the recommendation of dental floss. Studies available on the adjunct effect of flossing to adult brushing have short follow-up periods, only one older than 6 months (ROSEMA et al., 2008), and do not evaluate caries outcomes, dental calculus, loss of clinical insertion and quality of life. In addition, McGuire et al. (2014) recommend the incorporation of outcomes reported by the individual into clinical trials. Thus, randomized clinical trials that address these limitations are fundamental to evaluate the effectiveness of dental floss in the treatment of adult gingivitis.

METHODOLOGY This study will be a blinded randomized clinical trial. The sample will be composed of students from the Federal University of Santa Maria.

Eligible individuals who agree to participate in the study will sign the informed consent form.

This project was approved by the Ethics and Research Committee of the Federal University of Santa Maria (CAAE 53831716.5.0000.5346).

The calculated sample size was 76 individuals.

RANDOMIZATION Block randomization (10 units per block) will be performed. The randomization sequence will be generated by computer program (Random Allocation Software, version 1.0, May 2004). Concealment of randomization will be ensured by the use of opaque envelopes numbered from 1 to 76, which will correspond to the sequence from the first to the last participant to be randomized. Within each envelope will be the name of the experimental group that the individual will be allocated. A researcher (A.B.L.) not involved with outcome evaluations will be responsible for generating the sequence and maintaining concealment of randomization, and applying the interventions.

Individuals will be randomized into 2 groups according to whether or not they use dental floss:

* Group toothbrush (WITHOUT DENTAL FLOSS): Individuals will receive oral hygiene instructions with toothbrush only.
* Group toothbrush plus dental floss (DENTAL FLOSS): Individuals will receive oral hygiene instructions with toothbrush plusdental floss.

INTERVENTION The intervention consists of oral hygiene instructions with a toothbrush (WITHOUT DENTAL FLOSS) and toothbrush plus dental floss (DENTAL FLOSS), performed by a researcher (A.B.L.) not involved in the assessment of outcomes. The intervention will be performed within 8 weeks immediately after the baseline, corresponding to the efficacy study. Soon after this period, which will correspond to the effectiveness study, the interventions will not be repeated.

PERIODONTAL CLINICAL PARAMETERS Clinical parameters evaluated will be: Plaque Index (PL) (SILNESS; LÖE, 1964), Gingival Index (GB) (LÖE, 1967), plaque retentive factor (PRF), probing depth (PD), attachment level AL), bleeding probing (BOP), gingival recession (GR) and gingival crevicular fluid volume (GCFV).

Data will be analyzed using STATA 12.0 software (Stata Corporation, College Station, TX, USA). Descriptive analysis of PI, GB, GCFV and AL data will be performed using means, standard deviations and average percentage of sites with different IPI and GI scores. The differences in the mean PI, GB and GCFV over time between the groups and within the same group will be analyzed using the Poisson Multilevel Regression model.

The main outcome will be considered a reduction in gingival bleeding. The difference in the proportion of subjects who reached gingival health level after the interventions will be compared through the chi-square test with significance level of 5%. Adults with less than 15% of sites with gingival bleeding will be considered healthy (AMERICAN DENTAL ASSOCIATION, 2012). The unit of analysis will be the individual.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with at least 18 years of age, without loss of proximal clinical insertion, with papilla completely filling the interdental space and with at least 24 teeth will be eligible.

Individuals should present gingivitis in 15% of the proximal sites (gingival marginal bleeding, gingival index score 2, LÖE, 1967). Distal sites of the posterior teeth will not be counted in the analysis because they are not areas of flossing.

Exclusion Criteria:

* Dental students, individuals with xerostomia, pregnant women, diabetics, smokers, patients with orthodontic appliances and/or containment, individuals requiring antimicrobial prophylaxis to perform oral exams; who have used antibiotics/anti-inflammatories for the last three months and who have psychomotor disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-12-04 (Actual)

PRIMARY OUTCOMES:
gingival condition | 14 months
  The gingival condition will be assessed through the Gingival Index (GI) (Löe, 1967)

SECONDARY OUTCOMES:
Oral Health-related Quality of Life | 14 months
  The Health-related Quality of Life will be assessed through OHIP-14 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Carlos Heitor Cunha Moreira, Santa Maria, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reiniger APP, Cr Tavares R, Ortigara GB, Tatsch KF, Uliana JC, Wikesjo UM, Moreira CHC, Kantorski KZ. Effectiveness of dental floss in the management of gingival health: A 6-month follow-up of a randomized controlled clinical trial. Clin Oral Investig. 2024 May 16;28(6):319. doi: 10.1007/s00784-024-05693-4. PMID 38750375
- [Derived] Londero AB, Reiniger APP, Tavares RCR, Ferreira CM, Wikesjo UME, Kantorski KZ, Moreira CHC. Efficacy of dental floss in the management of gingival health: a randomized controlled clinical trial. Clin Oral Investig. 2022 Aug;26(8):5273-5280. doi: 10.1007/s00784-022-04495-w. Epub 2022 Apr 22. PMID 35451656